CLINICAL TRIAL: NCT02541201
Title: The Effect of the Consumption of Low-Fat Milk Enriched With Plant Sterols on Serum Low-Density Lipoprotein Cholesterol in Healthy Southern Chinese (COME-PASS)
Brief Title: The Effect of a Plant Sterols-Enriched Low-Fat Milk on Lipid Profile in Healthy Southern Chinese (COME-PASS)
Acronym: COME-PASS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Bernard Cheung, Sun Chieh Yeh Heart Foundation Professor in Cardiovascular Therapeutics, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CTC1430
Record Dates: First submitted 2015-08-26; First posted 2015-09-04 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Dyslipidemia
Keywords: Plant sterols; Low-Density Lipoprotein Cholesterol; Phytosterols
MeSH Terms: conditions — Dyslipidemias | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plant sterols-enriched low-fat milk (Experimental): Daily consumption of 1.5g of plant sterols as provided by two servings of 273 ml of plant sterols-enriched low-fat milk for consecutive 3 weeks, each serving taken right before breakfast and lunch.
  Interventions: Dietary Supplement: Plant sterols-enriched low-fat milk
- Low-fat milk (Placebo Comparator): Daily consumption of two servings of 273 ml of low-fat milk (without plant sterols) for consecutive 3 weeks, each serving taken right before breakfast and lunch.
  Interventions: Dietary Supplement: Low-fat milk

INTERVENTIONS:
Dietary Supplement: Plant sterols-enriched low-fat milk — The study product is a dried partly skimmed milk powder with no more than 12% milk fat (11.4g total fat/100g product) containing unesterified, unhydrogenated plant sterols.
  Arms: Plant sterols-enriched low-fat milk
Dietary Supplement: Low-fat milk — The placebo product is a dried partly skimmed milk powder.
  Arms: Low-fat milk

SUMMARY:
This is a randomized, double-blind, single-center, two-arm, placebo-controlled clinical trial that examine the effect of the consumption of a plant sterols-enriched low-fat milk. Half of the participants will consume of 1.5g of plant sterols daily as provided by two servings of the plant sterols-enriched low-fat milk product for 3 consecutive weeks, while the other half will consume placebo low-fat milk.

DETAILED DESCRIPTION:
Plant sterols are the naturally occurring functional equivalent of mammalian cholesterol. Plant sterols differ structurally from cholesterol by a methyl or ethyl group in their side chains and are not synthesized by the human body. These structural differences render them minimally absorbable in the intestine. It has been consistently reported that dietary incorporation of plant sterols(1.5-2 g/day) reduces serum low-density lipoprotein cholesterol (LDL-C) levels with minimal adverse events. The hypochoelsterolemic effects of plant sterols is explained by an inhibition of cholesterol absorption, which is ascribed to a competition with intestinal cholesterol for incorporation into mixed micelles, although other possible mechanistic explanation have been proposed.

ELIGIBILITY:
Inclusion Criteria:

* Southern Chinese male or female ≥ 18years.
* In good general health as evidenced by medical history
* Have the ability to understand the requirements of the study, provide written informed consent, including consent for the use and discloser of research-related health information, and comply with the study data collection procedures. Provide signed and dated informed consent form

Exclusion Criteria:

* Subject with familial hypercholesterolemia
* Ingestion of drugs known to interfere with lipid profiles, such as hormone replacement treatment, diuretics, beta-blockers, statin or other hypochoelsterolemic drug treatment
* Smoking > 10 cigarettes/day
* Subject with heavy alcohol intake (Alcohol > 3 glasses wine, or 2 beers, or 1 shot hard alcohol/day)
* Having milk intolerance or dislike
* Having major diseases such as diabetes (type I and type II), renal or liver diseases
* Subject presenting known allergy or hypersensitivity to milk proteins, soy and peanut
* Subject refusing to stop the consumption of plant sterols-enriched products if any during the study (other than the studied product)
* Subject receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters
* Subject currently involved in a clinical trial or in an exclusion period following participation in another clinical trial
* Pregnancy or lactation
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2015-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Mean of serum low-density lipoprotein cholesterol (LDL-C) | From baseline to week 3

SECONDARY OUTCOMES:
Change of serum LDL-C | From baseline to week 3
Change of high-density lipoprotein cholesterol (HDL-C) | From baseline to week 3
Change of total cholesterol | From baseline to week 3
Change of triglycerides (TAG) | From baseline to week 3
Change of serum creatinine | From baseline to week 3
Changes of fasting blood glucose | From baseline to week 3

CONTACTS AND LOCATIONS:
Overall Officials: Cheung Bernard Man Yung, Principal Investigator — Li Ka Shing Faculty of Medicine, The University of Hong Kong

REFERENCES:
- [Derived] Cheung CL, Ho DK, Sing CW, Tsoi MF, Cheng VK, Lee GK, Ho YN, Cheung BM. Randomized controlled trial of the effect of phytosterols-enriched low-fat milk on lipid profile in Chinese. Sci Rep. 2017 Jan 24;7:41084. doi: 10.1038/srep41084. PMID 28117400